CLINICAL TRIAL: NCT05322603
Title: Efficiency and Safety a Fixed Combination of Orphenadrine and Diclofenac for Postoperative Analgesia in Cardiac Surgery Patients
Brief Title: Efficiency and Safety a Fixed Combination of Orphenadrine and Diclofenac for Postoperative Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Petrovsky National Research Centre of Surgery (Other)
Responsible Party: Principal Investigator, Aleksandr Eremenko, Clinical Professor, Petrovsky National Research Centre of Surgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00191200
Record Dates: First submitted 2022-03-26; First posted 2022-04-12 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Analgesia
Keywords: analgesia, non-opioid, patient-controlled analgesia
MeSH Terms: conditions — Agnosia | interventions — Analgesics, Non-Narcotic; Diclofenac; Analgesics; Analgesia, Patient-Controlled

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the first group: a fixed combination of Orphenadrine and Diclofenac (Experimental): dynamics of points 100 mm visual-analog scale,minute inspiratory lung volume
  Interventions: Drug: Analgesics Non Opioid (Neodolpasse manufactured by Fresenius Kabi)
- the second group: patient-controlled analgesia (РСА) with Morphine (Experimental): dynamics of points 100 mm visual-analog scale,minute inspiratory lung volume
  Interventions: Drug: Analgesics

INTERVENTIONS:
Drug: Analgesics Non Opioid (Neodolpasse manufactured by Fresenius Kabi) — A decrease in the pain severity (VAS);opioid-sparing effect
  Other Names: Fixed combination of Orfenadrine and Diclofenac
  Arms: the first group: a fixed combination of Orphenadrine and Diclofenac
Drug: Analgesics — A decrease in the pain severity (VAS)
  Other Names: Patient-controlled analgesia (with Morphine)
  Arms: the second group: patient-controlled analgesia (РСА) with Morphine

SUMMARY:
The study will include 60 patients after cardiac surgery. The first group will include 30 patients who will use the drug Neodolpasse manufactured by Fresenius Kabi, which is a fixed combination of 30 mg of orphenadrine and 75 mg of diclofenac; the second group will consist of 30 patients who will use patient-controlled morphine analgesia (РСА) in the form of monotherapy.

DETAILED DESCRIPTION:
The patient signs an informed consent to participate in the study after tracheal extubation.The application of one or another method of influence is carried out by the method of random sampling (the envelope method). The drug Neodolpasse is used according to the following plan: in the form of an intravenous infusion of 250 ml for 2 hours 1 or 2 times a day with intervals between infusions about 12 hours. The second injection will be prescribed at VAS > 40 mm no earlier than 12 hours after the first. The first injection will begin immediately after tracheal extubation. Morphine analgesia controlled by the patient will begin 2 hours after tracheal extubation (the concentration of the drug will be 1 mg /ml; the initial or loading dose is 3 mg; the bolus dose was 1 mg; the lockout interval is 6 minutes; the 4-hour maximum dose is 10 mg; the rate of constant infusion is 0.1 mg / hour).

ELIGIBILITY:
Inclusion Criteria:

1. age from 18 years to 80 years inclusive
2. surgical access - median sternotomy
3. the first 2 hours after tracheal extubation
4. clear consciousness and productive contact with the patient
5. absence of erosive or ulcerative lesions of the mucous membrane of the esophagus, stomach and duodenum during preoperative esophago-gastro-duodenoscopy and clinical manifestations of gastrointestinal bleeding
6. no signs of renal dysfunction (KDIGO 0)
7. stable state of hemodynamics

Exclusion Criteria:

1. a history of mental illness
2. the presence of contraindications to the appointment of diclofenac and orphenadrine or individual intolerance to drugs of these groups
3. renal and hepatic insufficiency
4. perioperative brain lesions
5. postoperative bleeding>1.4 ml/kg/hour
6. severe cardiovascular (inotropic index>10) and/or respiratory (RaO2 /FiO2<200 mmHg) insufficiency

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-08-20 (Actual)

PRIMARY OUTCOMES:
visual-analog scale | hospitalisation period, an average of 24 hours
  dynamics of points 100 mm visual-analog scale

SECONDARY OUTCOMES:
the minute inspiratory lung volume using a spirometer | hospitalisation period, an average of 24 hours
  Comparison of minute inspiratory lung volume befor/after research using a spirometer
opioid-sparing effect | hospitalisation period, an average of 24 hours
  Comparison of the number of opioid analgesics
adverse events | hospitalisation period, an average of 1 week
  registration of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Alexander A. Eremenko, prof, Study Director — Head of the Intensive Care Unit; Lyubov S. Sorokina, Principal Investigator — anesthesiologist-resuscitator
Locations (1):
- Petrovsky Research National Centre of Surgery, Moscow, Russia